CLINICAL TRIAL: NCT03248063
Title: A Multicenter Non-inferiority Randomized Trial Comparing Cloxacillin Versus Cefazolin Efficacy for the Treatment of Bacteremia Caused by Methicillin-susceptible Staphylococcus Aureus (MSSA)
Brief Title: Non-inferiority Trial Comparing Cloxacillin vs Cefazolin in Methicillin-susceptible Staphylococcus Aureus Bacteremia
Acronym: CLOCEBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160943J
Record Dates: First submitted 2017-07-24; First posted 2017-08-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Bacteremia Due to Methicillin Susceptible Staphylococcus Aureus
Keywords: Staphylococcus aureus; bacteremia; cloxacillin; cefazolin
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia | interventions — Cloxacillin; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cloxacillin (Active Comparator): Intravenous treatment by cloxacillin, 25 to 50 mg/kg every 4 or 6 hours, without doing less than the minimum daily dose of 8 g/day and without exceeding the maximum daily dose of 12 g/day, administered as a 60-minutes infusion.
  Interventions: Drug: Cloxacillin
- Cefazolin (Experimental): Intravenous treatment by cefazolin, 25 to 50 mg/kg every 8 hours (without exceeding the maximum daily dose of 6 g/day), administered as a 30-minutes infusion.
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cloxacillin — Intravenous treatment by cloxacillin, 25 to 50 mg/kg every 4 or 6 hours, without doing less than the minimum daily dose of 8 g/day and without exceeding the maximum daily dose of 12 g/day, administered as a 60-minutes infusion. This treatment will be administered for at least 7 days by intravenous route.
  Dosing regimen will be adapted in patients with chronic renal failure (glomerular filtration rate below 30ml/min/1.73m²) and in patient with impaired hepatic function associated with renal impairment whatever the level of the estimation of the glomerular filtration rate, according to SPC.
  Arms: Cloxacillin
Drug: Cefazolin — Intravenous treatment by cefazolin, 25 to 50 mg/kg every 8 hours (without exceeding the maximum daily dose of 6 g/day), administered as a 30-minutes infusion. This treatment will be administered for 14 days by intravenous route. Dosing regimen will be adapted in case of glomerular filtration rate between 30-50ml/min according to SPC. As currently recommended, investigators will be encouraged to use the intravenous route for the entire duration of treatment. However, in order to interfere as little as possible with usual practice in each center, the antimicrobial therapy will be let to the choice of the physician in charge of the patient after a minimum of 7 days of intravenous treatment.
  Arms: Cefazolin

SUMMARY:
"Methicillin-susceptible Staphylococcus aureus (MSSA) bacteremia remains a major cause of community- or hospital-acquired bloodstream infections with an overall mortality estimated around 25%. Anti-staphylococcal penicillins (APs) such as oxacillin or cloxacillin are recommended as first-line agents. With the exception of first-generation cephalosporin (1GC) such as cefazolin, no alternative has yet proven a similar efficacy. Due to an unfavourable safety profile for high doses used in severe infection, an uneasy dosing schedule in patients with renal failure and possible recurrent stock-out events for APs, alternative to APs are needed. This led to propose an open-label, randomized, controlled parallel groups, phase IV, non-inferiority trial comparing the efficacy, the safety, and the ecological impact of cefazolin versus cloxacillin for the treatment of MSSA bacteremia in adults.

The primary objective is to compare the therapeutic efficacy of cefazolin vs cloxacillin at day 90 after the inclusion. "

DETAILED DESCRIPTION:
"Methicillin-susceptible Staphylococcus aureus (MSSA) bacteremia remains a major cause of community- or hospital-acquired bloodstream infections with an overall mortality estimated around 25%. Anti-staphylococcal penicillins (APs) such as oxacillin or cloxacillin are recommended as first-line agents. With the exception of first-generation cephalosporin (1GC) such as cefazolin, no alternative has yet proven a similar efficacy: studies evaluating other β-lactams exhibited 2 fold-increased rates of mortality, while a 3 fold-increased mortality rate was observed with vancomycin.

Recently, the safety of APs has been questioned, as both hypersensitivity reactions and renal impairment have been reported to be higher than 10%. Premature discontinuation of APs attributed to adverse events occurred in >20% of patients treated with high dosing of oxacillin (12g/day) for complicated MSSA bacteremia. This might be linked to the growing number of cumulative comorbid conditions and to ageing. In particular, administration and dosing schedule for APs are not well defined in patients with chronic kidney disease with decreased rate of glomerular filtration. Today, data are missing for renal adjustment.

In addition, stock-outs of essential antimicrobials are more and more frequent. In 2011, the production of the main generic for injectable oxacillin, distributed in France, was stopped. More recently, cloxacillin was also stock-out because of manufacturing problems. A limited production is currently available.

Due to an unfavourable safety profile for high doses used in severe infection, an uneasy dosing schedule in patients with renal failure and possible recurrent stock-out events for APs, alternative to APs are needed.

Cefazolin, intravenous 1GC, is more and more commonly used. Based on several large observational studies, its efficacy is believed to be similar to that of APs both in terms of relapse and mortality, even in complicated cases such as osteo-arthritis or infective endocarditis. The potential hydrolysis of cefazolin by Staphylococcus aureus type A ßlactamases had no clinical impact. These data led the American and European infectious disease Societies to consider cefazolin as the first alternative line agent for treatment of MSSA-associated infective endocarditis. Nevertheless, except for chronic dialysis question, all existing studies assessing the efficacy profiles of cefazolin compared to the APs contain a retrospective design and no randomized clinical trial (RCT) has been performed.

However, in the current context of growing bacterial resistance, especially for third-generation cephalosporins (3GCs) resistance in Enterobacteriaceae, the use of cefazolin, which has a large antibacterial spectrum, instead of APs, whose antibacterial spectrum is very narrow, remains to be investigated. Few data are available to assess the impact of cefazolin and APs on the bacterial floras.

This is an open-label, randomized, controlled parallel groups, phase IV, non-inferiority trial comparing the efficacy of cefazolin versus cloxacillin for the treatment of MSSA bacteremia in adults.

The primary objective is to compare the therapeutic efficacy of cefazolin vs cloxacillin at day 90 after the inclusion.

The primary endpoint is a composite efficacy criterion of (at least one of) the following:

* Survival at day 90
* Bacteriologic success at day 5
* Absence of relapse at day 90
* Clinical success at day 90.

Secondary objectives include, according to treatment group:

Efficacy objectives

1. To compare the mortality at day 90
2. To compare the bacteriological efficacy at day 3, at day 5 and at day 90
3. To compare the rate of bacteriologic relapse at day 90
4. To compare the clinical efficacy at day 7 and at day 90
5. To compare the proportions of patients for whom consensual treatment duration is respected Safety objectives
6. To compare the occurrence of any adverse event (AE) at day 7, at the end of studied antibiotic therapy (EoST) and at the end of all antibiotic therapy (EoAT)
7. To compare the occurrence of grade 3 or grade 4 AE at day 7, at EoST and at EoAT
8. To compare the rate of premature discontinuation of studied antibiotic therapy due to the occurrence of an adverse event
9. To compare the occurrence C. difficile infection

Ancillary studies will be performed for evaluating the impact of S. aureus beta lactamases on the effectiveness, for determination of PKPD (pharmacokinetic and pharmacodynamic) parameters of cloxacillin and cefazolin predictive of therapeutic effectiveness, and for comparing cloxacillin and cefazolin impact on the emergence of 3rd generation resistant enterobacteria and on the intestinal microbiota (evaluated by 16 rRNA (ribosomal ribonucleic acid) gene profiling).

Patients with a positive blood culture for Gram-positive cocci and a time-to-positivity ≤20 hours will be assessed for eligibility. The cut-off of 20 hours for the time-to-positivity was chosen according to data from the VIRSTA study, in which about 90% of SAB (staphylococcus aureus bacteremia) were positive in less than 20 hours after blood sampling. Median and 75th percentile were 13 hours and 18 hours after blood sampling. Concordant data have already been reported .

A rapid molecular test for detection of protein A, mecA and mecSCC genes will be performed on the blood culture by GeneXpert real-time PCR, according to the manufacturer's specifications (Cepheid, Sunnyvale, CA).

Patients with methicillin-susceptible Staphylococcus aureus positive blood culture will be randomized after full information and verification of inclusion criteria. Randomization will be stratified on center and vascular access-associated bacteremia with a 1:1 ratio.

There is no limitation on the nature of antibiotics that patients might receive prior to the randomization. However, antibiotic treatment active against MSSA should have begun in the last 48 hours before the randomization.

All patients will undergo transthoracic echocardiography within 7 days following randomization for diagnosing infective endocarditis. Other radiological exams will be performed depending on the clinical suspicion for the origin of bacteremia or for the presence of deep abscess.

According to the guidelines, patients with MSSA bacteremia will be treated with intravenous antimicrobial therapy for 2 weeks. The total treatment duration will be left to the choice of the clinician in charge of the patient but will be not below 14 days. Nevertheless, after 7 days, the nature of the antimicrobial treatment will be let to the choice of the clinician in charge of the patient. Treatment duration according to the final diagnosis will be defined by consensual guidelines. These guidelines are being developed using a methodology inspired by the Delphi method as part of the Tep-Star clinical trial. The coordinating investigator of the Tep-Star trial is Vincent Le Moing and its scientific director is Xavier Duval. Both are members of the scientific committee of this trial. Antimicrobials for switch of the first treatment line will be let to the choice of the investigator in charge of the patient.

Clinical evaluations for efficacy and safety will be performed at day -1, at day 7, at EoAT, and 90 days after the beginning of therapy. Blood cultures for efficacy evaluation will be performed at days 1, 3, 5 and 90. Biological evaluation for safety will be performed at days -1, 1, 3, 7, at EoST, at EoAT and at day 90.

The epidemiology of blaZ β-lactamases will be studied in all strains of S. aureus isolated from the blood culture vials.

The ancillary study of the antibiotic impact on the bacterial flora will be performed on a subgroup of 150 patients (75 in each treatment group). Rectal swabs will be collected just before and at day 7, at EoAT and at day 90.

The pharmacokinetic ancillary study will be performed on a subgroup of 50 patients (25 in each treatment group). For pharmacokinetic calculations, plasma cefazolin and cloxacillin levels will be determined at day 3, just before the 7th administration of cefazolin and the 9th administration of cloxacillin, and 1, 1.5, 2, and 4 hours after the beginning of infusion."

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Blood culture positive to MSSA identified by standard bacteriologic techniques or by GeneXpert PCR

Exclusion Criteria:

1. Previous type 1 or grade 3 - 4 according to CTCAE hypersensitivity reaction to beta-lactams
2. Known pregnancy or breastfeeding women
3. Parenteral antimicrobial therapy active against MSSA for more than 72 hours after the positive SA blood culture ponction
4. Chronic renal failure defined by a glomerular filtration rate estimated < 30 mL/min/1,73m².
5. Presence of an intra-vascular implant (vascular or valvular prosthesis or cardiovascular implantable electronic device)
6. Patient with implanted material considered to be infected by SAMS and whose antibiotic treatment is longer than 70 days
7. New cerebro-spinal signs in the preceding month
8. Clinical examination compatible with recent stroke (<1 month), brain abscess or meningitis
9. Current other antibiotic therapy which cannot be ceased or substituted by study treatment
10. Mixed blood culture with more than one pathogen (excluding contaminants: Corynebacterium sp., Propionibacterium sp., Coagulase-Negative Staphylococci)
11. coagulapthy with TP< 50% (excepted for patients under avk anticoagulant treatment)
12. Absence of written informed consent from the patient
13. Limitation of care with expected life duration below 90 days
14. Patient under guardianship or trusteeship
15. No affiliation to social security (beneficiary or assignee)
16. Subject already involved in another interventional clinical research evaluating a medicinal product

Secondary exclusion criteria:

1. Diagnosis of meningitis made after randomisation
2. Diagnosis of brain abscess made after randomisation
3. Diagnosis of multiple infection made after randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy | 90 days after beginning of antibiotic treatment
  "Composite efficacy criterion of the following:
  1. Survival at day 90
  2. Bacteriologic success at day 5
  3. Absence of relapse at day 90
  4. Clinical success at day 90"

SECONDARY OUTCOMES:
Mortality | day 90
  Mortality rate at day 90
Bacteriological efficacy | day 3, day 5 and day 90
  Proportions of patients with a negative set of blood culture at day 3, at day 5 and at day 90
Bacteriologic relapse | day 5
  Proportion of patients with bacteriologic success at day 5 in whom a strain of S. aureus with identical in vitro antibiotic susceptibility pattern than the one isolated at inclusion is isolated from at least 1 blood culture during the follow up
Clinical efficacy | day 7 and day 90
  Proportions of patients improving all signs and symptoms related to the infection at day 7 and at day 90
Proportions of patients for whom consensual treatment duration is respected | day 90
  Proportion of patients for whom the antibiotic duration from randomization is in accordance with consensual guidelines obtained by the Delphi method
Occurrence of any adverse event | at day 7 and up to 6 weeks
  Proportions of patients with any adverse event at day 7, at the end of studied antibiotic therapy (EoST) and at the end of all antibiotic therapy (EoAT)
Occurrence of grade 3 or grade 4 adverse event | at day 7 and up to 6 weeks
  7. Proportions of patients with any grade 3 or grade 4 adverse event at day 7, at EoST and at EoAT
Premature discontinuation of studied antibiotic therapy due to the occurrence of an adverse event | day 90
  Proportion of patients with premature discontinuation of studied antibiotic therapy due to the occurrence of an adverse event
Occurrence C. difficile infection | day 90
  Proportion of patients with C. difficile infection
Prevalence of BlaZ genes in S. aureus strains isolated from patients with MSSA bacteremia | at inclusion
  Proportion of type A, type B, type C and type D BlaZ genes
Link between BlaZ typing and bacteriologic efficacy | day 5
  Type of BlaZ gene. Proportion of patients with a negative blood culture at day 5.
MICs distribution of cefazolin and cloxacillin in S. aureus strains isolated from patients with MSSA bacteremia | at inclusion
  MICs of cefazolin and cloxacillin
Emergence of antimicrobial resistance in the faecal microbiota | at day 7, up to 6 weeks and at day 90
  Proportion of patients with emergence of 3rd generation cephalosporin-resistant Enterobacteriaceae in fecal swabs at day 7, at EoAT and at day 90
Changes in relative abundance of each bacterial phylum | at day 7, up to 6 weeks and at day 90
  comparison of the variation from baseline of the logarithm of proportions of each bacterial phylum at inclusion, EoAT and day 90
Changes in bacterial diversity within the intestinal microbiota | at day 7, up to 6 weeks and at day 90
  comparison of the change from baseline of shannon index within the intestinal microbiota between inclusion and day 90
Total body clearance of cloxacillin and cefazolin in patients with MSSA bacteremia | at day 3
Total body volume of distribution of cloxacillin and cefazolin in patients with MSSA bacteremia | at day 3
Area under the plasma concentration versus time curve (AUC) of cloxacillin and cefazolin | at day 5
Peak Plasma Concentration (Cmax) of cloxacillin and cefazolin | at day 5
Minimal inhibitory concentration (MIC) of cloxacillin and cefazolin | at day 5
Residual concentration (Cres) of cloxacillin and cefazolin | at day 5
The proportion of time between 2 administration during which the plasma concentration of the antimicrobial is above the MIC (%T>MIC). | at day 5

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Lescure, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- François-Xavier Lescure, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Burdet C, Saidani N, Dupieux C, Lemaignen A, Canoui E, Surgers L, Vareil MO, Lefort A, Lepeule R, Peiffer-Smadja N, Charmillon A, Le Moing V, Boutoille D, Tolsma V, Abgrall S, Wolff M, Tattevin P, Esposito-Farese M, Vandenesch F, Duval X, Tubiana S, Lescure FX; CloCeBa Study Group. Cloxacillin versus cefazolin for meticillin-susceptible Staphylococcus aureus bacteraemia (CloCeBa): a prospective, open-label, multicentre, non-inferiority, randomised clinical trial. Lancet. 2025 Nov 15;406(10517):2349-2359. doi: 10.1016/S0140-6736(25)01624-1. Epub 2025 Oct 17. PMID 41115439
- [Derived] Burdet C, Loubet P, Le Moing V, Vindrios W, Esposito-Farese M, Linard M, Ferry T, Massias L, Tattevin P, Wolff M, Vandenesch F, Grall N, Quintin C, Mentre F, Duval X, Lescure FX; CloCeBa study group. Efficacy of cloxacillin versus cefazolin for methicillin-susceptible Staphylococcus aureus bacteraemia (CloCeBa): study protocol for a randomised, controlled, non-inferiority trial. BMJ Open. 2018 Sep 1;8(8):e023151. doi: 10.1136/bmjopen-2018-023151. PMID 30173161